CLINICAL TRIAL: NCT01131234
Title: A Phase 1, Pharmacokinetic and Pharmacodynamic Study of the Combination of RO4929097 and Cediranib in Patients With Advanced Solid Tumors
Brief Title: Gamma-Secretase Inhibitor RO4929097 and Cediranib Maleate in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01428; NCI-2011-01428 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000673867; PJC-004 (Other: University Health Network-Princess Margaret Hospital); 8503 (Other: CTEP); U01CA132123 (NIH)
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-11

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Oligodendroglioma; Adult Brain Stem Glioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Adult Solid Neoplasm; Male Breast Carcinoma; Recurrent Adult Brain Neoplasm; Recurrent Breast Carcinoma; Recurrent Colon Carcinoma; Recurrent Melanoma; Recurrent Non-Small Cell Lung Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Ovarian Germ Cell Tumor; Recurrent Pancreatic Carcinoma; Recurrent Rectal Carcinoma; Recurrent Renal Cell Carcinoma; Stage III Pancreatic Cancer; Stage III Renal Cell Cancer; Stage IIIA Colon Cancer; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Ovarian Germ Cell Tumor; Stage IIIA Rectal Cancer; Stage IIIA Skin Melanoma; Stage IIIB Breast Cancer; Stage IIIB Colon Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Ovarian Germ Cell Tumor; Stage IIIB Rectal Cancer; Stage IIIB Skin Melanoma; Stage IIIC Breast Cancer; Stage IIIC Colon Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Ovarian Germ Cell Tumor; Stage IIIC Rectal Cancer; Stage IIIC Skin Melanoma; Stage IV Breast Cancer; Stage IV Non-Small Cell Lung Cancer; Stage IV Ovarian Cancer; Stage IV Ovarian Germ Cell Tumor; Stage IV Pancreatic Cancer; Stage IV Renal Cell Cancer; Stage IV Skin Melanoma; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Astrocytoma; Ependymoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Breast Neoplasms, Male; Brain Neoplasms; Breast Neoplasms; Colonic Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Carcinoma, Renal Cell | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (cediranib maleate and RO4929097) (Experimental): Patients receive gamma-secretase inhibitor RO4929097 PO QD on days 1-3, 8-10, and 15-17 (days 1-3, 8-10, 15-17 22-24, 29-31, and 36-38 of course 1 only) and cediranib maleate PO QD on days 1-21 (days 22-42 course 1 only). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: Gamma-Secretase Inhibitor RO4929097; Drug: Cediranib Maleate; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Gamma-Secretase Inhibitor RO4929097 — Given PO
  Other Names: RO4929097
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; Recentin
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I clinical trial is studying the side effects and best dose of giving gamma-secretase inhibitor RO4929097 and cediranib maleate together in treating patients with advanced solid tumors. Gamma-secretase inhibitor RO4929097 and cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Cediranib maleate also may stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the tolerability, maximum tolerated dose (equivalent to the recommended phase II dose), and safety profile of RO4929097 (gamma-secretase inhibitor RO4929097) in combination with cediranib (cediranib maleate) in patients with advanced malignancies.

SECONDARY OBJECTIVES:

I. To obtain pharmacokinetic (PK) profiles for RO4929097 when administered alone and for RO492907 and cediranib in combination, in order to evaluate for interactive effects in PK (if any) between these two agents.

II. To evaluate pharmacodynamic (PD) effects of RO492907 when administered alone and in combination, with the goal of identifying potential predictive and PD markers that need further exploration and validation in future trials.

III. To assess for preliminary antitumor efficacy of this drug combination, especially in breast cancer, malignant melanoma, colorectal cancer, pancreatic cancer, kidney cancer, high grade glioma, non-small-cell lung cancer, and ovarian cancer.

OUTLINE: This is a dose-escalation study.

Patients receive gamma-secretase inhibitor RO4929097 orally (PO) once daily (QD) on days 1-3, 8-10, and 15-17 (days 1-3, 8-10, 15-17 22-24, 29-31, and 36-38 of course 1) and cediranib maleate PO QD on days 1-21 (days 22-42 course 1 only). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Dose-escalation cohorts: Patients must have histologically and/or cytologically confirmed solid malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; expansion cohort: patients must have histologically and/or cytologically confirmed breast cancer, malignant melanoma, colorectal cancer, pancreatic cancer, kidney cancer, high grade glioma, non-small-cell lung cancer, or ovarian cancer
* Patients must have measurable or non-measurable disease; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan; measurable disease is not required to participate in this trial
* No limitation on prior therapy; however, there must be at least a 4 week interval between initiation of study treatment and any prior radiotherapy or systemic therapy, 6 weeks if the last regimen included carmustine (BCNU) or mitomycin C; exceptions may be made however, for low dose, non-myelosuppressive radiotherapy for symptomatic palliation; please contact the Princess Margaret Hospital (PMH) Phase I Consortium Central Office coordinator or the Principal Investigator if any questions arise about interpretation of this criterion
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3.0 x 10^9/L
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin >= 90 g/L (or >= 9 g/dL)
* International normalized ratio (INR) =< 1.3
* Total bilirubin normal =< institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x institutional upper limit of normal
* Serum creatinine < institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Left ventricular ejection fraction (LVEF) >= 50% by echocardiogram (ECHO)/multi gated acquisition scan (MUGA)
* Urine dipstick for protein of less than +1; for +1 or greater than +1 proteinuria on 2 consecutive dipsticks taken no longer than 1 week apart, 24-hour urine for protein is necessary and should be < 1 g/24 hours
* Patients must be able to swallow medication
* If women of childbearing potential do not abstain* from sexual activity they must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry; women of childbearing potential can either be abstinent or use two forms of contraception for the duration of study participation and for at least 12 months post-treatment; men must use condoms when sexually active with women for the duration of study participation and at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study and for 12 months after study participation, the patient should inform the treating physician immediately

  * Abstinent from sexual activity at least 4 weeks prior to study entry
  * Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of RO4929097 (serum or urine); a pregnancy test (serum or urine) will be administered every 3 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of RO4929097 and /or cediranib; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing RO4929097 and /or cediranib, the investigator must confirm and document the patient's use of two contraceptive methods or abstinence, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of RO4929097 and cediranib
  * Female patients of childbearing potential are defined as follows:

    * Patients with regular menses
    * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
    * Women who have had tubal ligation
  * Female patients may be considered to NOT be of childbearing potential for the following reasons:

    * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
    * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive months
    * Pre-pubertal females; the parent or guardian of young female patients who have not yet started menstruation should verify that menstruation has not begun; if a young female patient reaches menarche during the study, then she is to be considered as a woman of childbearing potential from that time forward
* Ability to understand and the willingness to sign a written informed consent document
* Archival tissue availability with consent for pharmacodynamic analysis is highly preferred but NOT an inclusion criterion

Exclusion Criteria:

* Patients who have had systemic therapy or radiotherapy or major surgery within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents within the past 30 days or have been previously treated with a gamma-secretase inhibitor and/or cediranib; exposure to other angiogenesis inhibitors (e.g. sorafenib, bevacizumab) is acceptable
* Patients with any meningeal metastases or untreated known brain metastases should be excluded from this clinical trial; patients with treated brain metastasis with radiologic and clinical evidence of stability, with no evidence of cavitation or hemorrhage in the brain lesions, are eligible providing that they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 1 week prior to randomization)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097 and/or cediranib used in the study
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible (except low dose warfarin for prophylaxis for central catheters)
* Patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) should be switched to alternative medications to minimize any potential risk; if such patients cannot be switched to alternative medications, they will be ineligible to participate in this study
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, active peptic ulcer disease, short gut syndrome, malabsorption syndrome of any type, total or partial bowel obstruction or inability to tolerate oral medications) that potentially impairs their ability to swallow or absorb are excluded
* Patients who are serologically positive for hepatitis A, B or C, or have a history of liver disease, other forms of hepatitis or cirrhosis are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study

  * Note: it is acceptable to use corrected calcium when interpreting calcium levels
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia other than chronic, stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with RO4929097 with or without cediranib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients with corrected QT interval (QTc) prolongation (defined as QTc interval >= 450 msec in males and 470 msec in females, by Bazett correction) or other significant electrocardiogram (ECG) abnormalities (i.e. clinically significant arrhythmias requiring medication or conduction delays such as 2nd or 3rd degree atrioventricular blocks, etc) are ineligible

  * History of risk factors for QT interval prolongation, including, but not limited to family or personal history of long QT syndrome, history of torsades de pointes, recurrent syncope without known etiology or sudden unexpected death
  * The need for antiarrhythmics or other concomitant medications with known potential to prolong QT interval
* Patients who have not recovered from side effects of previous systemic anticancer therapy to < Common Terminology Criteria for Adverse Events (CTCAE) grade 2 (except alopecia) prior to the first dose of combination
* Patients with a >= grade 2 diarrhea not under control with standard anti-diarrhea medications
* Patients with resting blood pressure (BP) consistently higher than, systolic > 150 mmHg and/or diastolic > 100 mmHg (in the presence or absence of a stable dose of anti-hypertensive medication) or poorly controlled hypertension, history of labile hypertension or poor compliance with anti-hypertensive medication

  * Blood pressure needs to be optimally controlled and < 150/100 for a period of at least 2 weeks prior to enrollment into the study
* Patients with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days of treatment
  * Any history of cerebrovascular accident (CVA) within the past 6 months
  * Prophylactic low-dose warfarin is permitted, but close monitoring of INR must be performed; baseline INR must meet the inclusion criteria; note: low molecular weight heparin is permitted
  * History of symptomatic cardiac dysfunction within the last 12 months including unstable angina, congestive heart failure (class III or IV heart failure as defined by the New York Heart Association [NYHA] functional classification system, myocardial infarction, cardiac angioplasty or stenting or bypass; patients with a significant cardiac history, even if controlled, should have a LVEF of >= 50% by ECHO or MUGA prior to study entry
* Patients previously treated with anthracyclines are eligible as long as their ejection fraction is > 50% by ECHO or MUGA prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of gamma-secretase inhibitor RO4929097 defined as the dose level at which < 1/6 patients experience dose-limiting toxicity as graded by the National Cancer Institute (NCI) CTCAE version 4.0 | 42 days
  Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest.
Incidence of adverse events as graded by the NCI CTCAE version 4.0 | Up to 4 weeks post-treatment
  Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest.

SECONDARY OUTCOMES:
PK profiles for both drugs | On days 1, 10, 22, and 38 of course 1, and then on day 1 of courses 2-6
  PK parameters will be calculated by non-compartmental methods.
PD effects of gamma-secretase inhibitor RO4929097 when administered alone and in combined with cediranib maleate | On days 1 and 22 of course 1 and on day 1 of course 2
  Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. Ninety-five percent confidence intervals will be provided for estimates of interest where possible.
Preliminary antitumor efficacy | Up to 4 weeks post-treatment
  Summary statistics, such as the mean, median, counts and proportion, will be used to describe patients' clinical characteristics. Objective response to treatment will be assessed using the RECIST criteria 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Hotte, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (2):
- Canada (2):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario